CLINICAL TRIAL: NCT07399652
Title: Artificial Intelligence-Guided Detection of Anatomical Markers to Enhance Safety in Third-Space Endoscopic Procedures
Brief Title: Artificial Intelligence-Guided Detection of Blood Vessels to Enhance Safety in Third-Space Endoscopic Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Abhishek Tyagi, Principal AI Engineer, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: AITSE-1
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Achalasia Cardia; Tumor
Keywords: Artificial Intelligence; Third Space Endoscopy; POEM; ESD; STER; EMR
MeSH Terms: conditions — Esophageal Achalasia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With Artificial Intelligence (Active Comparator): Endoscopist will see the AI generated segmentation mask
  Interventions: Device: AI generated segmentation mask for sub-mucosal blood vessels
- Without Artificial Intelligence (No Intervention): Endoscopist will not see the AI generated segmentation mask

INTERVENTIONS:
Device: AI generated segmentation mask for sub-mucosal blood vessels — Real time AI generated segmentation mask or delineation contours for sub-mucosal blood vessels visible on the endoscopy monitor.
  Arms: With Artificial Intelligence

SUMMARY:
This prospective study aims to evaluate the performance of a novel Artificial Intelligence (AI) clinical decision support tool during third space endoscopic procedures, such as Endoscopic Submucosal Dissection (ESD) and Peroral Endoscopic Myotomy (POEM).

While these procedures are effective for treating gastrointestinal neoplasms and motility disorders, they carry risks of intraprocedural bleeding and perforation if submucosal blood vessels are not correctly identified and coagulated. Building on previous retrospective validation, this study will assess whether a real-time artificial intelligence model can assist endoscopists in detecting and delineating blood vessels more accurately and faster during live human procedures.

DETAILED DESCRIPTION:
Background and Rationale

Third-space endoscopy procedures are technically demanding. The primary challenge lies in the inadvertent transection of submucosal vessels, which leads to bleeding that obscures the surgical field and increases the risk of perforation. Currently, vessel identification is entirely operator-dependent.

Our team has developed a deep-learning based artificial intelligence model trained on 250,000 annotated images from 150 POEM procedures. This model is optimized for minimal latency, allowing for real-time visual overlays (delineation) of blood vessels on the endoscopic monitor.

Study Objectives The primary objective is to evaluate the Vessel Detection Rate (VDR)-the proportion of vessels identified by the endoscopist when assisted by the AI compared to standard practice.

The study will also investigate:

Vessel Detection Time (VDT): The latency between a vessel appearing in the field of view and its identification.

Study Design & Workflow:

In this prospective study, the AI system will be integrated into the Olympus EVIS X1 series endoscopy stack. As the endoscopist navigates the submucosal space, the AI will provide real-time visual segmentation masks highlighting vessels. The performance will be recorded and compared against a post-procedure review by independent experts to calculate sensitivity and detection speed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Achalasia Cardia or neoplasms.

Exclusion Criteria:

* Patients with conditions deemed unsuitable for third space endoscopy procedures (e.g.: Candidiasis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Vessel Detection Rate (VDR) | 3 months
  the proportion of vessels identified by the endoscopist

SECONDARY OUTCOMES:
Vessel Detection Time (VDT) | 3 months
  The latency between a vessel appearing in the field of view and its identification.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Tyagi, Principal Investigator — Asian Intitute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scheppach MW, Mendel R, Muzalyova A, Rauber D, Probst A, Nagl S, Rommele C, Yip HC, Lau LHS, Golder SK, Schmidt A, Kouladouros K, Abdelhafez M, Walter BM, Meinikheim M, Chiu PWY, Palm C, Messmann H, Ebigbo A. Use of artificial intelligence in submucosal vessel detection during third-space endoscopy. Endoscopy. 2025 Jul;57(7):760-766. doi: 10.1055/a-2534-1164. Epub 2025 Feb 5. PMID 39909396
- [Result] Ebigbo A, Mendel R, Scheppach MW, Probst A, Shahidi N, Prinz F, Fleischmann C, Rommele C, Goelder SK, Braun G, Rauber D, Rueckert T, de Souza LA Jr, Papa J, Byrne M, Palm C, Messmann H. Vessel and tissue recognition during third-space endoscopy using a deep learning algorithm. Gut. 2022 Dec;71(12):2388-2390. doi: 10.1136/gutjnl-2021-326470. Epub 2022 Sep 15. PMID 36109151